CLINICAL TRIAL: NCT00796471
Title: A Comparative Evaluation of the Pharmacokinetics and Pharmacodynamics Under Fasting and Fed Conditions of 2 Paliperidone Extended-release Formulations With Paliperidone Oral Solution in Healthy Adults
Brief Title: A Pharmacokinetics and Pharmacodynamics Study Under Fasting and Fed Conditions With Paliperidone Extended-release and Immediate-release Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR004282
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mood Disorders; Antipsychotic drugs; Paliperidone ER
MeSH Terms: conditions — Schizophrenia; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of 2 extended-release (ER) formulations of 2 mg-eq paliperidone in comparison to the 2 mg immediate-release (IR) paliperidone oral solution and to evaluate the effect of food on the pharmacokinetics of these ER formulations. Additional objectives are to compare the pharmacodynamic effects (postural changes in blood pressure and heart rate), safety, and tolerability are to be evaluated in addition to exploring the relationship between CYP2D6 and CYP3A4/5genotype and paliperidone exposure.

DETAILED DESCRIPTION:
This study is designed as a single-center, open-label, randomized, 5 treatment-period, crossover study in healthy adults. The study consists of a screening phase and a treatment phase during which each volunteer will receive 5 treatments of study drug in a random order and separated by a washout period of at least 7 to 14 days. Treatments consist of a single oral dose of: A) paliperidone ER pellet formulation, (2 mg-eq) as 1 capsule of 2.5 mg, fasted; B) the same formulation as A but with food; C) paliperidone-coated ER OROS formulation (2 mg eq) as 2 tablets of 2 mg, fasted; D) the same formulation as C but with food; E) IR paliperidone oral solution, 2 mg (2 mL) of a 1 mg/mL solution, fasted. Alternative paliperidone ER formulations are being developed with the aim to increase the bioavailability without compromising the favorable effect on the orthostatic hypotension as seen with ER OROS paliperidone. Therefore, in this study, the pharmacokinetic and pharmacodynamic properties, as well as the effect of food, of 2 alternative paliperidone ER formulations using different mechanisms to achieve extended release of the drug will be investigated: a multiparticulate ER capsule formulation, containing coated pellets comprised of 3 coating layers, with both immediate and extended drug-release properties (pellet formulation; drug ratio extended- versus immediate-release layer: 9:1), and an OROS trilayer longitudinally compressed tablet formulation (Push-Pull delivery system) (overcoated-OROS formulation). Safety and tolerability will be monitored throughout the study. Single doses of paliperidone ER pellet formulation, (2 mg-eq) as 1 capsule of 2.5 mg, fasted; paliperidone ER pellet formulation, (2 mg-eq) as 1 capsule of 2.5 mg with food (high-fat breakfast); paliperidone-coated OROS ER formulation (2 mg-eq) as 2 tablets of 2 mg, fasted; paliperidone-coated OROS ER formulation (2 mg-eq) as 2 tablets of 2 mg with food (high-fat breakfast); IR paliperidone oral solution, 2 mg (2 mL) of a 1 mg/mL solution, fasted.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable weight as defined by body mass index (weight [kg]/height (m)²) range of 18.0 to 28.0 kg/m², inclusive
* Normotensive with supine (5 minutes) blood pressure between the range of 100 to 140 mmHg systolic, inclusive, and 60 to 90 mmHg diastolic, inclusive
* Healthy on the basis of a prestudy physical examination, medical history, electrocardiogram, and the laboratory results of blood biochemistry, hematology and urinalysis performed within 21 days before the first dose. If the results of the biochemistry, hematology or urinalysis testing are not within the laboratory's reference ranges the volunteer can be included only if the investigator judges that the deviations are not clinically significant. For liver function tests (alanine transaminase, aspartate transaminase, and bilirubin), the values must be contained within 2 times the upper limits of the normal laboratory reference ranges and for renal function tests, the values must be within the normal laboratory reference ranges
* Women must be postmenopausal for at least 1 year, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization and at the discretion of the investigator, total abstinence) before entry and throughout the study, as well as have a negative serum pregnancy test at screening. To ensure continued eligibility, women must have a negative urine test before each dose of study drug (Day -1 for each period).

Exclusion Criteria:

* Known allergy or history of significant hypersensitivity to heparin
* Recent history of alcohol or substance abuse. Test positive for the urine drug screen at screening or the urine drug screen or alcohol breath test at Day -1 for Period 1
* Relevant history of any cardiovascular, respiratory neuropsychiatric, renal, hepatic, gastrointestinal (including surgeries, and malabsorption problems), endocrine, or immunologic diseases
* A decrease of greater than or equal to 20 mmHg systolic blood pressure 3 minutes after standing, or with symptoms of lightheadedness, dizziness or fainting upon standing at screening
* Positive result for any of the serology tests (hepatitis B, C and HIV)
* History of smoking or use of nicotine-containing substances within the last 2 months, as determined by medical history and/or volunteer's verbal report. (Volunteers must agree to refrain from use throughout the study.)
* Drug allergy to risperidone, paliperidone, or any of its excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2003-06; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of 2 ER formulations of 2 mg-eq paliperidone in comparison with 2 mg IR paliperidone oral solution and to evaluate the effect of food on the pharmacokinetics of these ER formulations

SECONDARY OUTCOMES:
To compare the pharmacodynamic effects (postural changes in blood pressure and heart rate) of all treatments

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A pharmacokinetics and pharmacodynamics study under fasting and fed conditions with paliperidone extended-release and immediate-release formulations — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=579&filename=CR004282_CSR.pdf